CLINICAL TRIAL: NCT02761746
Title: Motivational Enhancement System for Adherence (MESA) for Youth Starting Antiretroviral Therapy (ART)
Brief Title: Motivational Enhancement System for Adherence (MESA) for Youth Starting ART
Acronym: MESA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wayne State University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Angulique Outlaw, Associate Professor, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 052115B3F; R01MH108442 (NIH)
Record Dates: First submitted 2016-02-29; First posted 2016-05-04 (Estimated); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Medication Adherence
Keywords: HIV; Adherence; Health Outcomes
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention Condition (MESA) (Experimental): MESA involves two sessions (ACASI assessment and intervention), one at study entry (prior to beginning ART) and one a month later. Then, participants will complete ACASI assessments only at 3, 6, 9, and 12 months. The first MESA session is tailored based on how important and how confident the person feels about taking medications as prescribed. The participant is also offered personalized feedback regarding immune status and HIV knowledge with actual adherence feedback provided in the second session. Finally, the participant may engage in goal setting. The second MESA session focuses on adherence behavior over the previous month and the consequences (good or bad) of that behavior.
  Interventions: Behavioral: MESA
- Control Condition (SH) (No Intervention): The SH control condition involves two sessions (ACASI assessment and control condition), one at study entry (prior to beginning ART) and one a month later. Then, participants will complete ACASI assessments only at 3, 6, 9, and 12 months. The first SH session targets healthy eating and physical activity and is matched for dose and length of time of the intervention session. Feedback and education are provided, if desired. Finally, the participants may engage in goal setting for healthy eating and physical activity. The second SH session focuses on the goals set during the first session and behavior over the previous month.

INTERVENTIONS:
Behavioral: MESA — MESA is tailored based on how important and how confident the participant feels about taking medications as prescribed. If the participant does not believe taking medications is important, they engage in a decisional balance exercise. If the participant believes taking medications is important, they move directly to confidence modules and goal setting. If the participant does not feel confident about taking medications, they engage in activities to boost self-efficacy. Participants are also offered personalized feedback regarding immune status and HIV knowledge with actual adherence feedback provided in the second session. Finally, goal setting is an option, and feedback regarding adherence behavior over the previous month.
  Arms: Intervention Condition (MESA)

SUMMARY:
This study is a multi-site (Detroit, MI; Los Angeles, CA; Philadelphia, PA, Washington, DC; Aurora, CO; Miami, FL; and Baltimore, MD), two-group randomized controlled trial testing a two-session intervention designed to increase motivation for adherence to antiretroviral treatment (ART) among youth living with HIV (YLH) newly recommended to begin medications. Participants are randomized to receive the intervention, Motivational Enhancement System for Adherence (MESA), or the control condition, System for Health (SH: healthy eating and physical activity information). Both groups receive the standard of care regarding the initiation of ART. ART adherence (visual analog scale and hair sample assay) and health outcomes (viral load results, and CD4 counts) are assessed. Additionally, potential mediators (HIV knowledge, motivation for adherence, and self-efficacy for adherence) and predictors of intervention response (substance abuse, mental health symptoms, executive functioning, and stressful life events) are assessed.

DETAILED DESCRIPTION:
Medication adherence rates among youth living with HIV (YLH) are inadequate to effectively manage the disease. Very few adherence interventions have been tested with youth, and those that have are difficult to implement in real-world settings due to high intensity of sessions or low attendance rates. Thus, there is a demand for innovative, feasible, and engaging behavioral interventions targeting adherence, especially among YLH, the largest initiators of antiretroviral treatment (ART). A universal primary prevention program is a novel approach to target adherence problems before they begin by providing a prevention intervention to all youth newly initiating ART. This study plans to test a brief, two-session, computer-delivered motivational intervention to prevent adherence difficulties among youth newly prescribed ART. All elements of the study (assessment, intervention, control condition) were piloted in a small multi-site randomized controlled trial (NIH-funded Adolescent Medicine Trials Medicine Network for HIV/AIDS Interventions: ATN). Results suggested feasibility and acceptability, as well as trends for improved adherence when comparing the intervention to an active control condition. For the proposed multi-site randomized clinical trial, youth newly beginning or restarting ART (N=200 from 7 ATN sites in the United States) will be randomize to the Motivational Enhancement System for Adherence (MESA) or to the control condition (System for Health: SH; nutrition and exercise information delivered by the same platform matched for dose). ART adherence (visual analog scale and hair specimen assays) and health outcomes (viral load results and CD4 counts) is the primary outcome. Potential mediators (HIV knowledge, motivation for adherence, and self-efficacy for adherence) on the treatment effects of MESA and moderators (substance abuse, mental health symptoms, executive functioning, and stressful life events) as predictors of differential intervention response will be assessed. It is hypothesized that participants randomized to MESA will show significantly greater adherence and health outcomes than participants randomized to SH over one year of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Youth living with HIV, ages 16 to 24 years 11 months, who are current patients at the 4 participating sites in Detroit, MI; Washington, DC; Los Angeles, CA; Philadelphia, PA; Aurora, CO; Miami, FL; and Baltimore, MD.
* Understands written and/or verbal English.
* Youth must have been verbally recommended to begin ART within the previous 12 weeks (recommendation could have first been made at an earlier time, but the youth must have been notified again by a health care provider in the previous 12 weeks), but has not been on ART for more than 30 days or verbally recommended to restart ART after being off ART for at least 6 months. Females who have received ART for the sole purpose of preventing maternal to child transmission in the past will be considered antiretroviral naïve.

Exclusion Criteria:

* Known pregnancy (pregnancy testing is not required).
* Inability to understand spoken or written English.
* Visibly distraught and/or visibly emotionally unstable (e.g., exhibiting suicidal, homicidal, manic or violent behavior).
* Active drug or alcohol use or dependence that, in the opinion of the site personnel, would interfere with ability to give true informed consent and to adhere to the study requirements.
* Active psychiatric condition that in the opinion of the site personnel, would interfere with the ability to give true informed consent and to adhere to the study requirements.
* Acute illness that, in the opinion of the treating clinician, would interfere with the participant's ability to adhere to the study requirements and/or interfere with the study objectives.
* Concurrent participation or participation within the previous 4 weeks, in any behavioral adherence intervention study or program.

Ages: 16 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 155 (Actual)
Dates: Start 2016-02-22 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Change in Medication Adherence (Visual Analog Scale) | 12 Months
  A change from baseline (1-month) medication adherence (Visual Analog Scale score) at 12 months via Audio-Computer Assisted Self-Interview (ACASI).
Change in Medication Adherence (Hair Sample Assay; physiological parameter) | 6 Months
  A change from baseline (6-month) medication adherence (hair sample collected from the head) at 12 months.
Change in Viral Load (biomedical measure) | 12 Months
  Viral load laboratory tests (biomedical measures of health status) will be collected, via a blood sample or obtained from medical record review, at baseline (6 weeks prior to enrollment) and 12-months. A change from baseline viral load at 12 months (decrease in viral load, increase undetectable status).
Change in CD4 count (biomedical measure) | 12 Months
  CD4 count laboratory tests (biomedical measures of health status) will be obtained from medical record review at baseline (6 weeks prior to enrollment) and 12-months. A change from baseline CD4 at 12 months (increase in the CD4 count).

SECONDARY OUTCOMES:
Information (HIV Treatment Knowledge score) as an intervention treatment effect | 12 Months
  Information, as measured by HIV Treatment Knowledge Score, will be obtained via ACASI at baseline, 1-month, and 3-, 6-, 9-, and 12-months.
Motivation (Readiness Ruler Importance score) as a intervention treatment effect | 12 Months
  Motivation, as measured by Rollnick's Readiness Ruler score adapted to focus on the importance of taking HIV medication will be obtained via ACASI at baseline, 1-month, and 3-, 6-, 9-, and 12-months.
Motivation (Decisional Balance for Adherence score) as a intervention treatment effect | 12 Months
  Motivation, as measured by the Decisional Balance for Adherence Score will be obtained via ACASI at baseline, 1-month, and 3-, 6-, 9-, and 12-months.
Behavioral Skills (Readiness Ruler Confidence score) as a intervention treatment effect | 12 Months
  Behavioral Skills, as measured by Rollnick's Readiness Ruler score adapted to focus on confidence for taking HIV medication, will be obtained via ACASI at baseline, 1-month, and 3-, 6-, 9-, and 12-months.
Behavioral Skills (Temptation Adherence score) as a intervention treatment effect | 12 Months
  Behavioral Skills, measured by the Temptation Adherence score, will be obtained via ACASI at baseline, 1-month, and 3-, 6-, 9-, and 12-months.
Predicting differential intervention response as measured by substance abuse (questionnaire score) | 12 Months
  Substance use, as measured by the Alcohol, Smoking, and Substance Involvement Screening Test v3.0: (ASSIST), will be obtained via ACASI at baseline, and 3-, 6- 9-, and 12-months.
Predicting differential intervention response as measured by executive functioning (questionnaire score) | 12 Months
  Executive functioning, as measured by the Behavior Rating Inventory of Executive Functioning-Adult Version: (BRIEF-A), will be obtained via ACASI at baseline, and 3-, 6- 9-, and 12-months.
Predicting differential intervention response as measured by structural barriers (questionnaire score) | 12 Months
  Structural barriers, as measured by the Services and Support score, will be obtained via ACASI at baseline, and 3-, 6- 9-, and 12-months.
Predicting differential intervention response as measured by mental health symptoms (questionnaire score) | 12 Months
  Mental health symptoms, as measured by the Brief Symptom Inventory-18: (BSI-18), will be obtained via ACASI at baseline, 1-month, and 3-, 6-, 9-, and 12-months.

CONTACTS AND LOCATIONS:
Overall Officials: Angulique Y Outlaw, PhD, Principal Investigator — Wayne State University; Sylvie Naar, PhD, Principal Investigator — University of Florida
Locations (7):
- United States (7):
  - Children's Hospital of Los Angeles, Los Angeles, California
  - University of Colorado School of Medicine, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Univeristy of Miami School of Medicine, Miami, Florida
  - Johns Hopkins School of Medicine, Baltimore, Maryland
  - Wayne State University, Detroit, Michigan
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Outlaw AY, Templin T, MacDonell K, Jones M, Secord E, Naar S. Motivational Enhancement System for Adherence for Adolescents and Young Adults Newly Recommended to Start Antiretroviral Therapy. J Acquir Immune Defic Syndr. 2025 Jan 1;98(1):49-56. doi: 10.1097/QAI.0000000000003530. PMID 39288943